CLINICAL TRIAL: NCT03495518
Title: Refinement and Early Evaluation of SPARK, an Approach to Enable Symptom Screening and Monitoring by Children Receiving Cancer Treatments
Brief Title: Enabling Symptom Identification and Tracking in Children Receiving Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Lillian Sung, Pediatric Oncologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB #1000053137
Record Dates: First submitted 2018-02-20; First posted 2018-04-12 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Pediatric Cancer; Quality of Life; Symptom Screening
Keywords: Cancer; Randomized Control Trial; Children; Hematopoietic stem cell transplantation; Quality of Life
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom feedback to Health Care Provider (Active Comparator): For those randomized to the intervention arm, symptom screening using SPARK will be completed once daily for 5 days on an iPad using the approach refined in aim 2. Daily SSPedi reports will be printed and provided in the patient chart. On days 1 and 3±1, a report describing symptoms that are "a lot" or "extremely" bothersome will be emailed to the physician providing direct medical care
  Interventions: Other: Symptom feedback to Health Care Provider
- Standard of care (Active Comparator): For those randomized to the control arm, a clinical research associate will visit the participant on days 1 and 5±1 and will obtain SSPedi scores on an iPad. Reports will not be printed or emailed to the physician.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Symptom feedback to Health Care Provider — These children will complete SPARK daily for 5 days in a row, daily symptom reports will be printed and provided in the patient chart. On days 1 and 3, a report describing symptoms that are "a lot" or "extremely" bothersome will be emailed to the physician providing direct medical
  Arms: Symptom feedback to Health Care Provider
Other: Standard of care — A clinical research associate will visit the participant on days 1 and 5±1 and will obtain SSPedi scores on an iPad. Reports will not be printed or emailed to the physician.
  Arms: Standard of care

SUMMARY:
Children with cancer and hematopoietic stem cell transplant (HSCT) recipients suffer from severe and bothersome symptoms because treatments are intense. So, the investigators developed SPARK (Supportive care Prioritization, Assessment and Recommendations for Kids), a website devoted to helping children track symptoms and providing a way to let doctors and nurses know which symptoms are bothersome. This study will examine the likelihood that children will complete SPARK once daily, help the investigators figure out how to improve the website so that children will use it, and help the investigators plan the large scale trial to test its efficacy in improving quality of life (QoL).

Participants will be children with cancer or HSCT recipients who are 8-18 years of age and who are expected to be in hospital or in clinic daily for 5 days.To determine the feasibility of a randomized controlled trial (RCT) of symptom feedback to healthcare providers

DETAILED DESCRIPTION:
Methods: Participants will be children with cancer or HSCT recipients who are 8-18 years of age and who can understand English, and who are expected to be in hospital or in clinic daily for 5 days.

SPARK RCT will be a pilot multi-center RCT in which we will randomize children to either undergo daily symptom screening for 5 days with symptom reports provided to the healthcare team or standard of care. Feasibility will be met if at least 30 participants are enrolled within one year and at least 75% complete at least 60% of evaluations.

Quality of the Idea Children receiving cancer treatment have excellent survival outcomes, in part, related to the provision of intensive therapies. Unfortunately, most children suffer and experience severe and bothersome treatment-related symptoms. Symptoms not only impact on QoL and morbidity but, in addition, may negatively influence future psychosocial functioning.

Symptoms remain unaddressed even during healthcare encounters because children do not complain and clinicians fail to ask about them. We recently developed SSPedi, a pediatric-specific symptom screening tool on an iPad. SSPedi, however, consists only of the questions which ask about symptoms. SPARK is the web-based application which will facilitate access to SSPedi, encourage symptom screening, generate reports and allow children to track their symptoms. Careful thought to design is required to ensure SPARK optimizes future use and has clinical utility. The proposed project output is a product that facilitates longitudinal symptom screening and provides the groundwork for a future RCT of symptom feedback.

ELIGIBILITY:
Inclusion Criteria:

* We will include children with cancer and HSCT recipients who are 8-18 years of age at enrollment and who can understand English.
* Participants may be inpatients or outpatients, and may be actively receiving cancer treatment or may have completed treatment.

Exclusion Criteria:

* Exclusion criteria will be illness severity, cognitive disability, or visual impairment that precludes utilization of SPARK according to the healthcare team.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of an RCT of symptom feedback to healthcare providers versus standard of care | Study will be enrolling for 1 year with a goal to enroll 30 participants. Feasibility will be determined once all 30 participants have completed the study after 1 year
  Will be determined by both the number of patients who are recruited for this study, and the number of patients who complete at least 60% of evaluations. We will aim to enroll 30 participants at SickKids over one year. Outcome feasibility will be met if at least 30 participants are enrolled within one year and at least 75% complete at least 60% of evaluations

SECONDARY OUTCOMES:
Pediatric Quality of Life (Peds QL) Cancer Module Acute Version | Measure will be completed by participant on day 5±1 day.
  Measures self-reported symptoms related to cancer treatment, capturing physical, psychological and cognitive health. 5-point likert scale ranging from 0(almost never) to 4 (almost always); there is no weighting of items. Scores are transformed on a scale from 0 to 100. Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Mean score is calculated= Sum of the items over the number of items answered.
  Total Score is used and calculated by: Sum of all the items over the number of items answered on all the Scales. Higher scores indicate lower problems.
Symptom Screening in Pediatrics (SSPedi) | Those randomized to the intervention arm measure will be completed by participant every day for 5 days. Those randomized to control arm measure will be completed by participant on Days 1 and 5±1 day.
  Self-reported symptom screening questionnaire asking pediatric patients (age 8-18) how bothered they are by 15 identified symptoms and side effects of cancer treatment. This 5-point Likert scale score from 0 (not bothered at all) to 4 (extremely bothered), and has a total score ranging from 0-60, with a higher number indicating more bother cancer-related symptoms. Likert scores will be summed for a total score that ranges from 0 (none) to 60 (worst possible).
Faces Pain Scale Revised | Measure will be completed on day 5±1 day.
  The Faces Pain Scale Revised is a self-report measure of pain intensity developed for children to score the sensation of pain on the 0-to-10 metric. The scale shows a close linear relationship with visual analog pain scale, counting left to right; 0" = "no pain" and "10" = "very much pain

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital For SickKids, Toronto, Ontario, Canada

DOCUMENTS (1):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT03495518/Prot_000.pdf